CLINICAL TRIAL: NCT04051892
Title: A Prospective, Open Label, Single Arm, Multicenter Study Evaluating the FixNip™ NRI Safety and Performance in Female Patients Seeking Reconstructive Surgery of the Nipple.
Brief Title: Multicenter Study Evaluating the FixNip™ NRI Safety and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FixNip Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLN003_0100
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Reconstruction of the Breast Nipple and Areola Complex

STUDY DESIGN:
Intervention Model Description: The sample size will be 10 female subjects undergoing reconstruction of the nipple, S/P breast reconstruction surgery as a result of breast cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation of FixNip™ NRI (Experimental): Female Patients Seeking Reconstructive Surgery of the Nipple
  Interventions: Device: FixNip™ NRI

INTERVENTIONS:
Device: FixNip™ NRI — The FixNip™ NRI is an implantable hypodermic, silicone implant specially designed for nipple areola definition

SUMMARY:
A prospective, Open Label, Single arm, Multicenter study Evaluating the FixNip™ NRI Safety and Performance in Female Patients Seeking Reconstructive Surgery of the Nipple.

DETAILED DESCRIPTION:
This is a Prospective, Open label, Single arm, Multicenter Study enrolling female patients with a history of breast cancer following breast conservation surgery or mastectomy with breast reconstruction, seeking reconstruction of the breast nipple and areola complex.

The study is designed to evaluate the long-term safety and performance of the FixNip NRI in patients undergoing nipple reconstruction procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 22-70 years.
* Patients of childbearing potential must agree to use methods of contraception and have negative pregnancy test at screening. Effective methods of contraception must be used throughout the study.
* History of breast cancer post mastectomy with breast implant or partial mastectomy (lumpectomy) of the central segment of the breast seeking reconstruction of the nipple and/or areola complex.
* At least 3 months post breast reconstruction surgery.
* Baker scale grade I or II capsular contracture.
* No evidence of any systemic or chronic disease that might influence wound healing and infection rate.
* Event free post breast and/or nipple reconstruction procedure, i.e. no skin infections or related infections that mandated antibiotic therapy, no wound dehiscence or any other related medical complications.
* Pinch test of intended nipple location on affected breast of at least 15 mm.
* Patient is willing to postpone tattooing until the end of follow-up period.
* Patient is willing and able to give their written informed consent.

Exclusion Criteria:

* Active malignant disease.
* Subject has a chronic disease or any medical status that, according to surgeon discretion, prohibits from inclusion in the study i.e. diabetes.
* History of tendency to produce hypertrophic scars or keloids.
* Current use of any medications that can interfere with wound healing, impair the immune system functionality, or impair blood clotting mechanisms.
* Active infection within the last 30 days.
* Pregnant or nursing women.
* Connective tissue disease.
* 'Lupus disease' defined as Systemic Lupus Erythematous or Discoid Lupus, or scleroderma defined as Progressive Systemic Sclerosis per history.
* Chronically treated with steroids or steroid therapy in a 3month period before surgery.
* Demonstrate psychological characteristics, which, in the opinion of the Investigator and/or consulting physician(s) are incompatible with the risks, involved with the surgical procedure, prosthesis and compliance with follow-up recommendations.
* Past or current capsular contracture defined as Baker III or IV.
* Participating in any other investigational study for either drug or device which can influence collection of valid data under this study.

Ages: 22 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Adverse event | 12 months
  Frequency and severity of Adverse Event . All adverse events occurring during the study will be reported

SECONDARY OUTCOMES:
Nipple Projection | 12 months
  Nipple projection in millimeter (mm)

OTHER OUTCOMES:
Satisfaction Evaluation | 12 months
  Rate of Patient satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scheflan, MD, Principal Investigator — Assuta MC; Ariel Tessone, MD, Study Director — Sheba MC
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel